CLINICAL TRIAL: NCT03431831
Title: Assessment of and Treatment Applied to Food Addiction to Encourage Self-Management of Obesity in a Rural Healthy Behaviors Clinic
Brief Title: Assessment of and Treatment Applied to Food Addiction in a Rural Healthy Behaviors Clinic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0763-16-FB
Record Dates: First submitted 2018-01-30; First posted 2018-02-13 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Counseling; bupropion hydrochloride, naltrexone hydrochoride drug combination; Pharmaceutical Preparations; Motivational Interviewing

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Statistician will make random assignment envelopes, clerical staff will collect intake forms and make envelope assignments according to randomization schedule. Participants will see different providers based on trial arm assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Intervention Control (Active Comparator): All participants will receive diet/physical intervention. One arm will receive diet/physical activity intervention alone as a Intervention/usual care condition.
  Interventions: Behavioral: Intervention Control
- Counselling (Experimental): These participants will receive usual care and counseling in the form of motivational interviewing weekly with goal setting for the first 5 weeks and monthly intervention for the final 5 months.
  Interventions: Behavioral: Intervention Control; Behavioral: Counselling
- Contrave (Experimental): These participants will receive usual care and prescription of Contrave for weight loss. They will be seen weekly for the first 5 weeks and monthly for the final 5 months.
  Interventions: Behavioral: Intervention Control; Drug: Contrave
- Contrave and counseling (Experimental): These participants will receive usual care of diet and physical activity recommendations and Contrave prescription and counseling (motivational interviewing interventions weekly for the first 5 weeks and then monthly for 5 months.
  Interventions: Behavioral: Intervention Control; Behavioral: Counselling; Drug: Contrave; Drug: Contrave and Counseling

INTERVENTIONS:
Behavioral: Intervention Control — diet recommendations of 1200 calorie limit for women daily and 1400 limit for men daily. Decreased foods that are high sugar, highly processed, low nutrient simple carbohydrates. Increased foods that are whole foods, lean proteins, complex carbohydrates and healthy fats. Switch from high calorie drinks to water for beverages.
Behavioral: Counselling — Usual care as listed in comparator intervention plus motivational interviewing to identify areas of barriers and how to overcome them, to help patient set achievable food, physical activity and beverage goals for themselves weekly and monthly. To identify whether knowledge or confidence counseling is more important for each participant and follow up with them. To help them learn self-management techniques for overeating.
  Arms: Contrave and counseling; Counselling
Drug: Contrave — In addition to usual care as described in the comparator intervention, these participants will be prescribed Contrave and raised to the therapeutic dosage within one month. They will be monitored closely for side effects and meds adjusted accordingly.
  Other Names: pharmaceutical
  Arms: Contrave; Contrave and counseling
Drug: Contrave and Counseling — This group of participants will receive a combination of all the above interventions including diet/physical activity prescription, motivational interviewing and Contrave.
  Other Names: motivational interviewing and pharmaceutical
  Arms: Contrave and counseling

SUMMARY:
Research purpose: The purpose of this pilot study is to assess obese clients for two phenotypes, those testing positive and those testing negative for Food Addiction (FA) (Yale Food Addiction Scale, YFAS) and determining the efficacy of four treatments: usual care (IC, dietary and physical activity instruction), individual motivational interviewing alone (MI), individual MI with pharmacotherapy (MI+P) for improving outcome measures within each phenotype, and pharmacological therapy (P).

Background/significance: Obesity has long been an epidemic in the U.S. and other countries. Numerous approaches have been tried to address obesity with limited success. The YFAS is a relatively new, validated instrument that can help researchers and practitioners assess obese clients for food addiction. Meeting the YFAS diagnosis criteria for FA suggests the need for a stronger intervention with close monitoring to assist these clients in self-management of their eating and physical activity behaviors.

Proposed methods/approach: The investigators propose assessing obese clients with the YFAS as part of their intake once they are referred to the Healthy Behaviors Clinic by Regional West physicians/practitioners. A nurse researcher with expertise in MI and a nurse practitioner will perform intake assessments, obtain consent and randomly assign participants in each phenotype (positive or negative for FA) to one of three treatment groups (usual care, individual MI alone, and individual MI with pharmacotherapy). Interventions will occur over 6 months. A clinical psychologist with expertise in the YFAS (University of Michigan) will serve as a consultant on this project and a registered dietitian (University of NebraskaLincoln) will serve as a co-investigator.

Expected outcomes: The investigators expect that MI and MI+P and P will be more effective in improving outcome measures than IC. We also expect that response to the treatments will differ between the two obesity phenotypes (those testing positive and those testing negative for FA).

DETAILED DESCRIPTION:
Treatment Assignment:

Both treatment groups,Those who test positive for and those who test negative for FA (food addiction) will be assigned to one of four treatment arms, IC, MI, MI/P and P. All will receive dietary and exercise information.

After consenting, each participant be administered the YFAS to determine their obesity phenotype (positive or negative for FA). Participants within each phenotype will be randomly assigned to one of the intervention (MI or MI+P, or P) or the IC information control (diet and physical activity instruction, which will be no less than current standard of care) treatment groups using a randomization schedule (assignments in numbered, sealed, opaque envelopes; one set for each phenotype) 1:1:1:1 ratio, provided by our statistician, Dr. Struwe. Phenotype assessment and treatment assignment will continue until the sample size (n=10) is met for each phenotype-treatment group category. Those participants in the control group will be seen at the same time periods as each treatment group to maintain their interaction time with the clinic. Participants will receive diet and exercise instruction at each time point.

Intervention Conditions (MI, MI+P):

MI is theorized to decrease a patients ambivalence and increase his/her perceived behavioral control (self-efficacy) for limiting highly processed and high in fat and sugar foods (HPFS) and increasing complex carbohydrates (CC) intake by emphasizing personal choice and control in decision-making and by affirming the patients self-management ability. Interventionist nurses will deliver MI sessions following data collection at baseline,1, 2,3, and 4 weeks and 2, 3, 4, 5, and 6 months to promote sustained behavioral change.50 A written MI algorithm will be used to ensure uniform implementation of the intervention.

MI will be operationalized by the nurse asking the patient about his/her knowledge , limiting HPFS/increasing CC and natural fat intake, defining FA, and explaining why it is important to limit their HPFS/increase their CC and natural fat intake. The nurse will ask the patient to rate the importance of limiting HPFS/increasing CC and natural fat intake (scale of 1-10) and their confidence in their ability to do so (scale of 1-10). The nurse will focus on the lower score and ask the patient why they chose that score and what they thought it would take to increase the number. If the patient rates the importance of understanding of limiting HPFS/increasing CC and natural fat intake low, the nurse will provide information on the benefits of limiting HPFS/increasing CC and natural fat intake to reduce the their risk of obesity, diabetes, heart disease, and numerous other co-morbidities associated with overweight. If the patient rates their confidence in their ability to limit HPFS/increase CC and natural fat intake as low, the nurse will provide the patient with strategies to decrease barriers and increase confidence, such as a list of healthy snack food choices, stepped changes (3 sodas per day to 2 sodas and 1 water per day, etc.), and having the patient choose healthy foods at the store. The same questions will be asked at each time point. Nurse responses will be tailored to the specific motivational issues of each individual patient at each time point. During each session, the nurse will document the patients responses to the MI algorithm (levels of confidence, importance, and readiness to change), their perceived barriers and concerns, and suggestions to address them/setting achievable goals. The MI documentation form will ensure that all nurses collect the same data and provides a record that the nurses can reference during their sessions to help them adjust each MI session to the patients individual needs. If a participant reveals a new barrier that is not included in the training materials, the nurses will meet with team members to discuss the new barrier and strategies to address it will be shared with all interventionists.

In the group with pharmacotherapy added to the MI, the naltrexone-buproprion (Contrave) protocol will be added to the patients intervention. Dosing protocols will be followed for treatment of obesity: Orally, 1 tablet (90mg/8mg) initially week 1; increase by 1 tablet/day each subsequent week until daily maintenance dose of 2 tablets twice daily (360 mg bupropion/32 mg naltrexone) is achieved at the start of week 4. Use will be discontinued at month 4 if no clinical response is observed. This drug (Contrave) is to be taken with a high fat meal.

In the pharmacotherapy group alone, Dosing protocols will be followed for treatment of obesity: Orally, 1 tablet (90mg/8mg) initially week 1; increase by 1 tablet/day each subsequent week until daily maintenance dose of 2 tablets twice daily (360 mg bupropion/32 mg naltrexone) is achieved at the start of week 4. Use will be discontinued at month 4 if no clinical response is observed. This drug (Contrave) is to be taken with a high fat meal.

IC Information Control Condition:

The IC control group will receive diet and physical activity information to encourage them to adopt healthier eating (limit HPFS/increase CC intake) and physical activity behaviors. IC information sessions will occur at the same time points as the intervention sessions (baseline, 1, 2,3, and 4 weeks and 2, 3, 4, 5, and 6 months) and will be similar in length. The PI and co-PIs will develop information packets for each session, (self-management, avoiding highly processed low-nutrient simple carbohydrates (LNSC) foods, low intensity physical activity, avoiding highly processed fatty foods, medium intensity physical activity, avoiding LNSC beverages, importance of water as a beverage to hydrate and reduce cravings, avoiding high fat beverages, high intensity physical activity, importance of CC intake).

Data Collection:

All research personnel will be Collaborative Institutional Training Initiative (CITI Program)-trained. A nursing student will assist the nurse researchers with data collection. Each data collector will undergo fidelity checks (performed by the PI) for each measurement procedure before they will be allowed to collect data. They will also be trained in using the ASA24-2016® dietary recall, so they can assist the patients as needed.

Outcome Measures:

YFAS: (Gearhardt et al, 2009; 2013). The current version of the YFAS, the YFAS 2.0, will be used to assess participants obesity phenotype (positive or negative for FA). This measures adapts the eleven DSM-5 diagnostic criteria for substance-related and addictive disorders when the substance is HPFS foods. In order to meet the diagnostic threshold on the YFAS, individuals must report at least two of the eleven diagnostic indicators of FA plus clinically significant impairment or distress.

Automated Self-Administered 24-hour Recall, version ASA24-2016®:

The Automated Self-Administered 24-hour Recall, version ASA24-2016® (National Cancer Institute, http://epi.grants.cancer.gov/asa24) will be completed at each time point to assess changes in patients dietary intake. This web-based 24 hour dietary recall instrument has been used effectively by hundreds of researchers and has face validity and similar intake results to the AMP.10 A strength of the ASA24-2016® is that it includes most traditional American foods/ingredients (Thompson, 2015).

Height: The participants height will be used in determining BMI and BIA measures. We will use the average of 2 heights (cm) measured with the Seca EC0123 stadiometer. During measurement, patients will be in socked feet with heels placed against the back of the platform and facing straight forward.

Body Composition: Bioelectrical impedance analysis (BIA) will be used to determine body composition. Estimated standard error for BIA is ± 3.5-5%, (American College of Sports Medicine, 2009). The investigators will use a Tanita SC-250 body composition analyzer and follow a standardized protocol to measure percent body fat, body fat mass, fat free mass, percent body water, muscle mass, bone mass, BMI, and visceral fat. The software also classifies patients as underfat, healthy, overfat, or obese based on percent body fat, age and gender.

Waist circumference: The investigators will use the average of 2 measurements (cm) performed with the patient standing erect with their arms at their sides. Waist circumference will be measured at the uppermost lateral border of the right ilium at the end of normal expiration using an inelastic tape measure positioned around the trunk parallel to the floor. This measure is included because it is a better indicator of body fat and, therefore, health risk than BMI(Griffiths, 2012). In addition, results of a recent study in this population demonstrated that waist circumference has potential as a means of identifying patients with or at risk for obesity and hypertension (Aguirre, 2015).

Blood Pressure: The investigators will use the average of 2 blood pressure measurements performed using an Omron HEM- 907 automatic blood pressure monitor. The measurements will be performed while the patient is quiet and still using the appropriate sized cuff placed snugly around the upper arm approximately 2 to 3 cm above the antecubital fossa with the mark on the cuff aligned with the artery.

Determinants of Change Measures:

MI Algorithm Questions: These reflect the Predicting and Changing Behavior Theory (PCBT) determinants of behavior change (the patients perceptions toward limiting HPFS/increasing CC intake). They assess patient attitudes/beliefs (importance score), perceived norms (perceived barriers), and perceived behavioral control/self-efficacy (confidence score). These measures will be recorded by the interventionist nurses during each MI session for their assigned patients.

If a subject experiences success in managing their weight while participating in the study,(which will be determined by a 5% decrease in BMI or body fat or total body mass over 4 months) the subject may continue with the weight management plan after completing all study related visits.

All participants may continue with clinic visits following the study and may have available to them, usual care, MI, Contrave (unless they have taken it in the study and it was not effective), and bariatric surgery options.

All subjects taking Contrave will be screened at each visit for suicidal ideation. In addition, they will be asked to call Dr. Bowman immediately if they have any such feelings or symptoms of suicidal ideation. If they present with suicidal ideation, Dr. Bowman will interview them using the Suicide Screening Algorithm (see documents) to determine the severity of the symptoms and make additional medical referrals as necessary. If the case is emergent, they will be immediately escorted to the ER or asked to come into the ER, if it is a phone visit. . If the case is urgent, they will be referred to psychiatric personnel in the office where Dr. Bowman practices as a Psychiatric Nurse Practioner. They will be withdrawn from the study at this time and Dr. Aguirre will be notified. Dr. Bowman will follow up with these patients.

At the six month visit a PHQ-9 and the YFAS (from the WALI) will be readministered. An appt for a 12 month sustainability measure will be set up.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/Obese Adult patients (age 19 years -65)
* eligible based on WALI screening tool

Exclusion Criteria:

* Inability to understand and read English.
* Women pregnant or lactating.
* persons with terminal illness

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trina M Aguirre, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Regional West Medical Center-University of Nebraska Medical Center, Scottsbluff, Nebraska
  - Regional West Physicians Clinic, Scottsbluff, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koehler A, Aguirre T, Schulte E, Bowman R, Struwe L. Secondary analysis of YFAS 2.0 symptom counts, impairment/distress, and food addiction severity in adults with overweight/obesity. Eat Weight Disord. 2021 Oct;26(7):2393-2399. doi: 10.1007/s40519-020-01077-1. Epub 2021 Jan 3. PMID 33389719

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Additional persons enrolled to replace withdrawals.
Groups:
- FA+ Intervention Control; FA- Intervention Control: All participants will receive diet/physical intervention. One arm will receive diet/physical activity intervention alone as a Intervention/usual care condition.
  Intervention Control: diet recommendations of 1200 calorie limit for women daily and 1400 limit for men daily. Decreased foods that are high sugar, highly processed, low nutrient simple carbohydrates. Increased foods that are whole foods, lean proteins, complex carbohydrates and healthy fats. Switch from high calorie drinks to water for beverages.
- FA+ Counselling; FA- Counseling: These participants will receive usual care and counseling in the form of motivational interviewing weekly with goal setting for the first 5 weeks and monthly intervention for the final 5 months.
  Intervention Control: diet recommendations of 1200 calorie limit for women daily and 1400 limit for men daily. Decreased foods that are high sugar, highly processed, low nutrient simple carbohydrates. Increased foods that are whole foods, lean proteins, complex carbohydrates and healthy fats. Switch from high calorie drinks to water for beverages.
  Counselling: Usual care as listed in comparator intervention plus motivational interviewing to identify areas of barriers and how to overcome them, to help patient set achievable food, physical activity and beverage goals for themselves weekly and monthly. To identify whether knowledge or confidence counseling is more important for each participant and follow up with them. To help them learn self-management techniques for overeating.
- FA+ Contrave; FA-Contrave: These participants will receive usual care and prescription of Contrave for weight loss. They will be seen weekly for the first 5 weeks and monthly for the final 5 months.
  Intervention Control: diet recommendations of 1200 calorie limit for women daily and 1400 limit for men daily. Decreased foods that are high sugar, highly processed, low nutrient simple carbohydrates. Increased foods that are whole foods, lean proteins, complex carbohydrates and healthy fats. Switch from high calorie drinks to water for beverages.
  Contrave: In addition to usual care as described in the comparator intervention, these participants will be prescribed Contrave and raised to the therapeutic dosage within one month. They will be monitored closely for side effects and meds adjusted accordingly.
- FA+ Contrave and Counseling; FA- Contrave and Counseling: These participants will receive usual care of diet and physical activity recommendations and Contrave prescription and counseling (motivational interviewing interventions weekly for the first 5 weeks and then monthly for 5 months.
  Intervention Control: diet recommendations of 1200 calorie limit for women daily and 1400 limit for men daily. Decreased foods that are high sugar, highly processed, low nutrient simple carbohydrates. Increased foods that are whole foods, lean proteins, complex carbohydrates and healthy fats. Switch from high calorie drinks to water for beverages.
  Counselling: Usual care as listed in comparator intervention plus motivational interviewing to identify areas of barriers and how to overcome them, to help patient set achievable food, physical activity and beverage goals for themselves weekly and monthly. To identify whether knowledge or confidence counseling is more important for each participant and follow up with them. To help them learn self-management techniques for overeating.
  Contrave: In addition to usual care as described in the comparator intervention, these participants will be prescribed Contrave and raised to the therapeutic dosage within one month. They will be monitored closely for side effects and meds adjusted accordingly.
  Contrave and Counseling: This group of participants will receive a combination of all the above interventions including diet/physical activity prescription, motivational interviewing and Contrave.
Period: Overall Study
Arm/Group | FA+ Intervention Control | FA+ Counselling | FA+ Contrave | FA+ Contrave and Counseling | FA- Intervention Control | FA- Counseling | FA-Contrave | FA- Contrave and Counseling
Started | 8 | 10 | 10 | 10 | 13 | 14 | 11 | 10
Completed | 6 | 8 | 8 | 9 | 9 | 10 | 10 | 9
Not Completed | 2 | 2 | 2 | 1 | 4 | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FA+ Intervention Control | FA+ Counselling | FA+ Contrave | FA+ Contrave and Counseling | FA- Intervention Control | FA- Counseling | FA-Contrave | FA- Contrave and Counseling | Total
Number analyzed (Participants) | 8 | 10 | 10 | 10 | 13 | 14 | 11 | 10 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 10 | 10 | 13 | 14 | 11 | 10 | 86
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 10 | 8 | 12 | 13 | 9 | 9 | 78
  Male | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 1 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 7 | 7 | 10 | 8 | 10 | 6 | 10 | 7 | 65
  Ethnicity: Hispanic | 1 | 3 | 0 | 2 | 3 | 6 | 1 | 3 | 19
  Ethnicity: Native American | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 10 | 10 | 13 | 14 | 11 | 10 | 86
Weight in lbs [Mean (Full Range); unit: Weight in Kilograms] | 231.9 [159.8 to 298] | 272.9 [180.8 to 362.6] | 221.7 [177.8 to 275.0] | 274.9 [179.8 to 411.8] | 250.5 [145.8 to 348.0] | 213.1 [133.4 to 351.6] | 242.9 [189.0 to 357.2] | 201.9 [160.8 to 319.4] | 238.7 [133.4 to 411.8]
Body Mass Index (BMI) in Kilograms/m2 [Mean (Full Range); unit: Kilograms/m2] | 39 [28.7 to 51.5] | 42.1 [30.6 to 55.1] | 39.9 [31.5 to 50.1] | 40.7 [30.9 to 63.0] | 35.5 [24.7 to 53.2] | 35.2 [25.9 to 64.7] | 38.7 [30.8 to 53.1] | 35 [26.9 to 53.2] | 38.3 [24.7 to 64.7]

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Weight in lbs
Time Frame: difference between baseline and 6 months
Population: difference between first and last weight measure among each group
Measure: Mean (Full Range); unit: lbs
Arm/Group | FA+ Intervention Control | FA+ Counselling | FA+ Contrave | FA+ Contrave and Counseling | FA- Intervention Control | FA- Counseling | FA-Contrave | FA- Contrave and Counseling
Number analyzed (Participants) | 6 | 8 | 8 | 9 | 9 | 10 | 10 | 9
lbs | -2.08 [-8.7 to 4.7] | -3.42 [-10.6 to 3.2] | -4.36 [-7.5 to 3.6] | -2.4 [-10.4 to 4.4] | -0.2 [-7.1 to 5.9] | -2.5 [-9.1 to 4.3] | -3.3 [-9.6 to 1.8] | -2.74 [-10.2 to 6.9]

2. Primary Outcome: Body Mass Index (BMI)
Description: Body Mass Index (BMI): Underweight Below 18.5, Normal 18.5-24.9, Overweight 25.0-29.9, Obesity 30.0 and Above
Time Frame: difference between baseline and 6 months
Population: difference between first and last BMI measure among each group
Measure: Mean (Full Range); unit: kg/m2
Arm/Group | FA+ Intervention Control | FA+ Counselling | FA+ Contrave | FA+ Contrave and Counseling | FA- Intervention Control | FA- Counseling | FA-Contrave | FA- Contrave and Counseling
Number analyzed (Participants) | 6 | 8 | 8 | 9 | 9 | 10 | 10 | 9
kg/m2 | -0.87 [-3.4 to 1.8] | -1.36 [-3.6 to 1] | -0.63 [-2.8 to 1.3] | -0.97 [-2.5 to 1.4] | -0.1 [-2.3 to 2.3] | -1.1 [-3.4 to 1.4] | -1.26 [-3.5 to 0.2] | -1.22 [-3.8 to 1.9]

ADVERSE EVENTS:
Time Frame: 18 months from baseline
Groups:
- Intervention Control/ FA-; Intervention Control/FA +: All participants will receive diet/physical intervention. One arm will receive diet/physical activity intervention alone as a Intervention/usual care condition.
  Intervention Control: diet recommendations of 1200 calorie limit for women daily and 1400 limit for men daily. Decreased foods that are high sugar, highly processed, low nutrient simple carbohydrates. Increased foods that are whole foods, lean proteins, complex carbohydrates and healthy fats. Switch from high calorie drinks to water for beverages.
- Counselling/ FA-; Counseling/FA+: These participants will receive usual care and counseling in the form of motivational interviewing weekly with goal setting for the first 5 weeks and monthly intervention for the final 5 months.
  Intervention Control: diet recommendations of 1200 calorie limit for women daily and 1400 limit for men daily. Decreased foods that are high sugar, highly processed, low nutrient simple carbohydrates. Increased foods that are whole foods, lean proteins, complex carbohydrates and healthy fats. Switch from high calorie drinks to water for beverages.
  Counselling: Usual care as listed in comparator intervention plus motivational interviewing to identify areas of barriers and how to overcome them, to help patient set achievable food, physical activity and beverage goals for themselves weekly and monthly. To identify whether knowledge or confidence counseling is more important for each participant and follow up with them. To help them learn self-management techniques for overeating.
- Contrave/FA-; Contrave/FA+: These participants will receive usual care and prescription of Contrave for weight loss. They will be seen weekly for the first 5 weeks and monthly for the final 5 months.
  Intervention Control: diet recommendations of 1200 calorie limit for women daily and 1400 limit for men daily. Decreased foods that are high sugar, highly processed, low nutrient simple carbohydrates. Increased foods that are whole foods, lean proteins, complex carbohydrates and healthy fats. Switch from high calorie drinks to water for beverages.
  Contrave: In addition to usual care as described in the comparator intervention, these participants will be prescribed Contrave and raised to the therapeutic dosage within one month. They will be monitored closely for side effects and meds adjusted accordingly.
- Contrave and Counseling/FA-; Contrave and Counseling/FA+: These participants will receive usual care of diet and physical activity recommendations and Contrave prescription and counseling (motivational interviewing interventions weekly for the first 5 weeks and then monthly for 5 months.
  Intervention Control: diet recommendations of 1200 calorie limit for women daily and 1400 limit for men daily. Decreased foods that are high sugar, highly processed, low nutrient simple carbohydrates. Increased foods that are whole foods, lean proteins, complex carbohydrates and healthy fats. Switch from high calorie drinks to water for beverages.
  Counselling: Usual care as listed in comparator intervention plus motivational interviewing to identify areas of barriers and how to overcome them, to help patient set achievable food, physical activity and beverage goals for themselves weekly and monthly. To identify whether knowledge or confidence counseling is more important for each participant and follow up with them. To help them learn self-management techniques for overeating.
  Contrave: In addition to usual care as described in the comparator intervention, these participants will be prescribed Contrave and raised to the therapeutic dosage within one month. They will be monitored closely for side effects and meds adjusted accordingly.
  Contrave and Counseling: This group of participants will receive a combination of all the above interventions including diet/physical activity prescription, motivational interviewing and Contrave.
Arm/Group | Intervention Control/ FA- | Counselling/ FA- | Contrave/FA- | Contrave and Counseling/FA- | Intervention Control/FA + | Counseling/FA+ | Contrave/FA+ | Contrave and Counseling/FA+
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/11 | 0/10 | 0/8 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/11 | 0/10 | 0/8 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14 | 0/11 | 0/10 | 0/8 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT03431831/Prot_SAP_002.pdf